CLINICAL TRIAL: NCT06204549
Title: Impact du Bilan et de la Prise en Charge Des comorbidités en médecine Interne Sur le Risque Cardiovasculaire
Brief Title: Impact of Assessment and Management of Comorbidities in Internal Medicine on Cardiovascular Risk
Acronym: COMMEDCARDIO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL22_0390; 2023-A00012-43 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-05

CONDITIONS: Adverse Cardiac Event; Major Adverse Cardiac Events
Keywords: Cardiovascular Risk; Comorbidities
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Comorbidities screening and management (Other)
  Interventions: Other: Screening and management of cormobidities

INTERVENTIONS:
Other: Screening and management of cormobidities — During the routine care assessment and as part of the research, patients will :
  * Fill in cardiovascular risk assessment score: Life's simple 7
  * Provide an additional blood sample (1 dry tube of 7 mL and 1 heparin tube of 7 mL) during their biological testing. These samples will be used for lipoprotein (a) testing and biological collection.
  After hospital discharge, patients will be contacted by telephone at 3 and 12 months for re-evaluation and will fill in the Life's simple 7 score. Prior to this contact, patients will have biological tests as prescribed just before hospital discharge (including blood ionogram, creatinine, liver assessment, lipid assessment (LDL, HDL, triglycerides), fasting blood sugar test, A1C test, urinary albumin/creatinine ratio, protein/ urinary creatinine ratio). They will weigh themselves and take blood pressure self-measurements over 3 days.

SUMMARY:
The aim of assessing and managing cardiovascular risk is to avoid, limit or delay cardiovascular morbidity and mortality. Planned internal medicine hospitalization is developed around the management of cardiovascular risk in patients at high cardiovascular risk, whether in primary prevention or secondary prevention.

During planned hospitalization, patients benefit from comprehensive, personalized and adapted care for their comorbidities and their CVRF (cardiovascular risk factors).

This study will make it possible to evaluate this overall course of multidisciplinary management of comorbidities of patients at high cardiovascular risk.

DETAILED DESCRIPTION:
The aim of assessing and managing cardiovascular risk is to avoid, limit or delay cardiovascular morbidity and mortality. Planned internal medicine is developed around the management of cardiovascular risk in patients at high cardiovascular risk, whether in primary prevention patients, combining several cardiovascular risk factors CVRF (arterial hypertension, metabolic syndrome, diabetes, dyslipidemia, etc.), or patients in secondary prevention who have several CVRFs and have already had a major cardiovascular event such as ischemic heart disease, heart failure.

During scheduled hospitalization, patients benefit from comprehensive care. Additional examinations include measurement of blood pressure, cardiac ultrasound, vascular Dopplers, usual biological assessment (lipid, glycemic, renal, iron assessment, CRP), and on a case-by-case basis, ventilatory polygraphy to screen for obstructive sleep apnea hypopnea syndrome, pulmonary function tests if the patient is a smoker to screen for chronic obstructive pulmonary disease, coronary function test to screen for ischemic heart disease if indicated. Comorbidities are thus identified and summarized, and patients benefit from personalized and adapted care for their comorbidities and CVRFs.

Cardiovascular risk reduction strategy programs targeting high-risk patients are essential and their evaluation is necessary.This study will make it possible to evaluate this overall course of multidisciplinary management of comorbidities in patients at high cardiovascular risk in internal medicine.

The innovative nature of the project is the possibility to cross-reference the comorbidities and the cardiovascular and metabolic data of these patients at high cardiovascular risk with their evolving risk level over time. This will also make it possible to highlight which markers are the most effective to better stratify cardiovascular risk, or even consider personalized phenotyping. The coexistence of all these parameters within the same database represents a unique opportunity to study their respective influences in a population of patients at high cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* High-Risk Cardiovascular patients either receiving:

  * Primary prevention because they have never had a cardiovascular event but have several cardiovascular risk factors such as high blood pressure particularly resistant, metabolic syndrome, diabetes , dyslipidemia, metabolic steatosis
  * Or secondary prevention because they have already had a major cardiovascular event such as ischemic heart disease, heart failure
* Aged 18 and over
* Patient benefiting from comorbidities assessment during their planned hospitalization in the internal medicine department.

Exclusion Criteria:

* Patient refusal
* Subject not registered in social security system
* Pregnant or breastfeeding woman
* Patient unable to give their informed consent, protected adult, vulnerable people
* Subject deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2027-05-21 (Estimated); Study Completion 2027-11-21 (Estimated)

PRIMARY OUTCOMES:
Screening and management of comorbidities effect on cardiovascular risk factors | 3 months after enrollment
  Effect of comorbidities screening and management on cardiovascular risk factors in patients at high-risk of a cardiovascular event.
  The life's simple 7 score will be used at enrollment and 3 months afterward. The score includes four modifiable behaviors (smoking, weight, healthy/unhealthy eating diet and physical activity) and three biometric measures (blood pressure, cholesterol and blood sugar level). These seven factors are classified into three categories: ideal, intermediate and poor. Life's Simple 7 summary score ranges from 0 to a maximum of 14 points, with a higher score indicating healthier status.

SECONDARY OUTCOMES:
Screening and management of comorbidities effect on cardiovascular risk factors | 12 months after enrollment
  Effect of comorbidities screening and management on cardiovascular risk factors in patients at high-risk of a cardiovascular event.
  The life's simple 7 score will be used at 12 months after enrollment. The score includes four modifiable behaviors (smoking, weight, healthy/unhealthy eating diet and physical activity) and three biometric measures (blood pressure, cholesterol and blood sugar level). These seven factors are classified into three categories: ideal, intermediate and poor. Life's Simple 7 summary score ranges from 0 to a maximum of 14 points, with a higher score indicating healthier status.
Screening and management of comorbidities effect on blood pressure | 3 and 12 months after enrollment
  Effect of comorbidities screening and management on the evolution of cardiovascular risk factor "blood pressure" 3 and 12 months after hospital discharge compared to hospitalization.
  Measurement method: Holter blood pressure measurement during hospitalization, and self-measured blood pressure average over 3 days at 3 and 12 months after hospitalization using cuff device for self-measurement.
Screening and management of comorbidities effect on patient's weight | 3 and 12 months after enrollment
  Effect of comorbidities screening and management on the evolution of cardiovascular risk factor "weight" at 3 and 12 months after hospital discharge compared to hospitalization.
  The patient's weight will be measured using a weighing scale.
Screening and management of comorbidities effect on the balance of cholesterol | 3 and 12 months after enrollment
  Effect of comorbidities screening and management on cardiovascular risk factor "cholesterol" by evaluating the evolution at 3 and 12 months after hospital discharge compared to hospitalization of biological tests: HDL (high-density lipoprotein), LDL(low-density lipoprotein) and triglycerides.
Screening and management of comorbidities effect on tobacco consumption | 3 and 12 months after enrollment
  Effect of comorbidities screening and management on the evolution of cardiovascular risk factor "tobacco consumption" (weaned or still acive,level of consumption) at 3 and 12 months after hospital discharge compared to hospitalization.
Screening and management of comorbidities effect on the balance of blood sugar level | 3 and 12 months after enrollment
  Effect of comorbidities screening and management on cardiovascular risk factor "blood sugar" by evaluating the evolution of fasting blood sugar test results at 3 and 12 months after hospital discharge compared to hospitalization.
Screening and management of comorbidities effect on A1C level | 3 and 12 months after enrollment
  Effect of comorbidities screening and management on the evolution of A1C test results at 3 and 12 months after hospital discharge compared to hospitalization in diabetic patients.
Cardivascular events incidence | 12 months after enrollment
  Description of the incidence of cardiovascular events including cardiovascular mortality.
Initial participant's comorbidities | At enrollment
  Exploration of demographic characteristics and initial comorbidities as factors associated with the evolution of cardiovascular risk factors and markers, for cardiovascular risk stratification purpose.
  Charlson Comorbidity Index (CCI) will be used at enrollment.The Index assesses comorbidity level by taking into account both the number and severity of 19 pre-defined comorbid conditions. It provides a weighted score of a patient's comorbidities which can be used to predict short term and long-term outcomes such as function, hospital length of stay and mortality rates.The total score in the CCI is derived by summing the assigned weights of all comorbid conditions presented by the patient. Higher scores indicate a more severe condition and consequently, a worse prognosis.
C-reactive protein levels | At enrollment
  Exploration of C-reactive protein (CRP) levels as an associated factor with the evolution of cardiovascular risk markers for cardiovascular risk stratification purpose
Lipoprotein a levels | At enrollment
  Exploration of Lipoprotein a levels as an associated factor with the evolution of cardiovascular risk factors and markers for cardiovascular risk stratification purpose.

CONTACTS AND LOCATIONS:
Overall Officials: Camille ROUBILLE, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University Hospital, Montpellier, France